CLINICAL TRIAL: NCT03398824
Title: Pilot Study of Metformin for Patients With Fanconi Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Akiko Shimamura, Director, Bone Marrow Failure and Myelodysplastic Syndrome Program, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00026540
Record Dates: First submitted 2017-12-13; First posted 2018-01-16 (Actual); Results first posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Fanconi Anemia
Keywords: Fanconi Anemia; Metformin
MeSH Terms: conditions — Fanconi Anemia | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental): Receive metformin HCl
  Interventions: Drug: metformin HCl

INTERVENTIONS:
Drug: metformin HCl — Receive metformin HCl

SUMMARY:
This is a single institution, open-label, single arm pilot study of Metformin in patients with Fanconi Anemia (FA) and cytopenias with the primary endpoint of hematologic response. This study will also assess safety, tolerability, and the biologic effects of Metformin in patients with FA.

ELIGIBILITY:
Inclusion Criteria:

* Age > 6 years and ≤35 years
* Lansky/Karnofsky performance status ≥ 50% for patients ≥16 years of age and Lansky ≥ 50% for patients <16 years of age (see Appendix A)
* Diagnosis requirement
* Participants must have a clinical diagnosis of Fanconi Anemia.

  * Participants must have confirmed diepoxybutane-mitomycin C (DEB/MMC) stress testing to document diagnosis of Fanconi Anemia.
  * Patients must have at least one of the following cytopenias: Hemoglobin <10g/dL; Platelets <100k/uL; Absolute neutrophil count <1000/uL
* Participants must have normal organ function as defined below:

  * Hepatic Function : Total bilirubin ≤ 1.5 x upper limit of normal for age; alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≤ 135 U/L
  * Renal Function: A serum creatinine based on age/gender as follows:

Age Maximum Serum Creatinine (mg/dL) Male Female

1. to < 2 years 0.6 0.6
2. to < 6 years 0.8 0.8

6 to < 10 years 1 1 10 to < 13 years 1.2 1.2 13 to < 16 years 1.5 1.4

≥ 16 years 1.7 1.4

AND

• Creatinine clearance ≥ 60 mL/min/1.73 m2 for participants with creatinine levels above institutional normal

* Normal cardiac status as documented clinically, otherwise they will need an echocardiogram prior to enrollment
* Serum bicarbonate must be >17.
* Participants of child-bearing or child-fathering potential must agree to use adequate contraception (hormonal birth control; intrauterine device; double barrier method; or total abstinence) throughout their participation, including up until 30 days after last dose of Metformin.
* Patients must be able to swallow pills.
* Ability to understand and/or the willingness of the patient (or parent or legally authorized representative, if minor) to provide informed consent, documented using an institutionally approved informed consent procedure

Exclusion Criteria:

* Patients must not have undergone prior bone marrow transplantation.
* Patients must not have very severe aplastic anemia at the time of enrollment which would require bone marrow transplantation (as defined by at least 2 out of the following 3: Absolute Neutrophil Count (ANC) <200k/uL, platelets <20k/uL, absolute reticulocyte count <40k/uL).
* Patients must not be taking any other concurrent medications to improve their hematopoiesis such as androgens or growth factors such as Granulocyte colony-stimulating factor (G-CSF), erythropoietin (EPO), or thrombopoietin (TPO) mimetics. There is a one month wash-out period for prior therapies including androgens.
* Pregnant participants will not be entered on this study given that the effects of Metformin on the developing human fetus are unknown.
* Breastfeeding mothers are not eligible because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Metformin.
* Patients must not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to Metformin.
* Patients must not have uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients must not have prior history of symptomatic hypoglycemia over the past year or hypoglycemia with glucose <50mg/dL on screening and baseline laboratory assessments.
* Patients must not have type 1 diabetes mellitus.
* Patients must abstain from alcohol as part of this study.
* Patients must not have a diagnosis of myelodysplastic syndrome or leukemia, or other concurrent malignancy undergoing treatment.
* Patients must not have vitamin B12 deficiency.
* Patients must not have Glucose-6-Phosphate Dehydrogenase (G6PD) deficiency.

Ages: 6 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2020-10-09 (Actual); Study Completion 2020-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Akiko Shimamura, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pollard JA, Furutani E, Liu S, Esrick E, Cohen LE, Bledsoe J, Liu CW, Lu K, de Haro MJR, Surralles J, Malsch M, Kuniholm A, Galvin A, Armant M, Kim AS, Ballotti K, Moreau L, Zhou Y, Babushok D, Boulad F, Carroll C, Hartung H, Hont A, Nakano T, Olson T, Sze SG, Thompson AA, Wlodarski MW, Gu X, Libermann TA, D'Andrea A, Grompe M, Weller E, Shimamura A. Metformin for treatment of cytopenias in children and young adults with Fanconi anemia. Blood Adv. 2022 Jun 28;6(12):3803-3811. doi: 10.1182/bloodadvances.2021006490. PMID 35500223

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Arm
Started | 14
Completed | 12
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 9.4 [6.0 to 26.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Hematologic Response
Description: Hematologic response is defined by specific increases in erythroid, platelet, and neutrophil counts.
  Erythroid response: Hemoglobin (Hgb) increase by >1.5g/dL for non-transfusion dependent patients and for patients who are transfusion dependent: Transfusion independence Only transfusions given for Hgb ≤8g/dL or for symptoms will be counted in the response evaluation
  Platelet response: If initially <20k/uL to start, then must increase to >20k/UL with an absolute increase of 100%. If initially ≥20k/uL to start, then must have an absolute increase of >30k/UL
  Neutrophil response: If initially <500/uL to start, then must increase to >500/uL with an absolute increase of > 250/uL. If initially ≥500/uL to start, then must have an absolute increase of >500/uL
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 14
Participants | 4
Statistical Analysis 1: Comparison: Treatment Arm; Test type: Other — Fanconi Anemia is a rare disease. Therefore, the primary end point of the study was to assess the proportion of subjects with a HR during 6 months of metformin treatment; sample size was calculated assuming that a HR rate < 20% suggests preliminary efficacy of treatment that warranted additional investigation and, conversely, that the study should be deemed futile if the rate of HR was <5%; response rate = 30.8, 90% CI 2-sided [11.3 to 57.3]; Fanconi Anemia is a rare disease. Therefore, the primary end point of the study was to assess the proportion of subjects with a HR during 6 months of metformin treatment; sample size was calculated assuming that a HR rate >20% suggests preliminary efficacy of treatment that warranted additional investigation and, conversely, that the study should be deemed futile if the rate of HR was <5%

ADVERSE EVENTS:
Time Frame: Study enrollment through 30 days after completion of treatment, up to 7 months
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 12/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (N=14)
Diarrhea (Gastrointestinal disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-02-28): https://cdn.clinicaltrials.gov/large-docs/24/NCT03398824/Prot_SAP_ICF_001.pdf